CLINICAL TRIAL: NCT01267474
Title: Reducing the Use and the Consumption of Sugar by School Lunch Cooks in Public Schools: a Cluster Randomized Trial
Brief Title: Reducing the Use of Sugar by School Lunch Cooks in Public Schools
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rio de Janeiro State University (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Rio de Janeiro State University, Rio de Janeiro State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNPQ:474135/2006-3
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-11

CONDITIONS: Sugar Intake
Keywords: School children; Sugar intake; Nutritional education program
MeSH Terms: interventions — Sugars

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional education (Experimental)
  Interventions: Other: Nutritional education
- Control (No Intervention)
  Interventions: Other: Control

INTERVENTIONS:
Other: Nutritional education — A nutritional education program was carried out during seven months of one school year aiming to reduce added sugar in school meals by the school lunch cooks and in their own consumption.
  All women in the intervention group participated in three sections about sugar consumption and one section on food labeling, as well as recipes competition of with reducing sugar.
  Printed material and gifts, such as mugs, refrigerator magnets and small purses with the logo of the campaign were given to the participants.
  All sections of education were delivered in the schools. The activities required 20 to 30 minutes and were facilitated by trained research assistants. Printed instructions and orientations on the facilitation process supported the assistants' efforts.
  Other Names: Use and consumption of sugar; School lunch cooks
  Arms: Nutritional education
Other: Control — The control group received only three one-hour general sessions on health issues.
  Other Names: General sessions on health issues
  Arms: Control

SUMMARY:
The main objective was to evaluate the effect of a nutritional education program for school lunch cooks, aiming to reduce added sugar in schools meals and in their sugar intake.

DETAILED DESCRIPTION:
Although Brazil is the largest producer and one of the world's largest consumers of sugar, research on sugar consumption is still a weak point among health indicators and there are no population studies to investigate the sugar intake in Brazilian population. Available data have shown reduction in the consumption of refined sugar (-37% between 1996 and 2003) but significant increase in consumption of soft drinks (400%), which constitute the main vehicle for consumption of added sugar. Moreover, studies have shown the adverse effects of excessive consumption of added sugar in dental caries and health, as excess energy intake hence in weight gain. Although several factors are associated with weight gain in adolescents, adults and elders, and several strategies have been released by both Brazil and International Agencies, as the Global Strategy, increased weight gain, particularly in adolescents, has been observed in several countries with large increase in Brazil, justifying specific projects to evaluate which messages, strategies and proposals for intervention would be effective.

ELIGIBILITY:
Inclusion Criteria:

* Women who were working in the function of school lunch cook in the schools.

Exclusion Criteria:

* Pregnancy, male.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2007-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Sugar intake | 10 months
  Reducing added sugar in the schools meals by school lunch cooks and in their sugar intake.

CONTACTS AND LOCATIONS:
Overall Officials: Rosely Sichieri, PhD, Principal Investigator — Rio de Janeiro State University
Locations (1):
- Rio de Janeiro State University, Rio de Janeiro, Rio de Janeiro, Brazil